CLINICAL TRIAL: NCT03267641
Title: A Multi-National Cohort Study On The Impact Of Intra-Tumoural Genomic Heterogeneity And The Immune Micro-Environment On The Clinical Trajectory Of Resected Hepatocellular Carcinoma
Brief Title: Prospective Cohort Study on the Clinical Trajectory of Resected Hepatocellular Carcinoma
Acronym: PLANET
Status: Completed | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: AHCC07
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Intra-tumour heterogeneity; Cancer immunotherapy; Tumour microenvironment; Driver mutations; Precision Medicine
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour samples Blood samples Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatocellular carcinoma (HCC) is the 6th most common cancer in the world but the 2nd most important cause of cancer death. Because of its highly heterogeneous nature, the current approach to identifying druggable targets have not delivered efficacious therapies in HCC and is a main reason for the high case fatality. Even when surgical resection is potentially curative in early disease, tumor recurrence remains high and long term survival poor because of the absence of useful adjuvant therapy.

To address these unmet needs, the investigators bring together internationally recognized scientists from genomics and immunology and established clinician investigators in a synergistic team. This TCR capitalizes on recent collaborative advances made by the PIs in the consortium. The investigators have shown through multi-region sampling of freshly resected HCC and phylogenetic analysis, that significant intra-tumoral heterogeneity exists and have identified the specific positions of known clonal drivers. Simultaneously the investigators have analyzed the immune landscape of the tumor microenvironment with deep immune-phenotyping and found unique inter-patient immune landscapes predictive of clinical trajectory.

This TCR is a prospective study that samples resected HCC from multi-ethnic sites within the established Asia-Pacific Hepatocellular Carcinoma (AHCC) Trials Group, which has enrolled approximately 1000 patients through 6 multi-center trials in 35 centers in the region. Clinical trajectories are tracked and genomic and immunological studies are repeated when tumors recu r, to confirm clonally dominant driver mutations and immunological processes that are targetable. Concurrently, representative pre-clinical models will be developed from the tissues sampled.

The investigators aim to combine these approaches to overcome the challenges posed by genomic heterogeneity and to guide the development of therapeutics and precision medicine in HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients, 21 to 80 years of age at the time of signature of the informed consent form.
2. Histologically proven HCC after liver resection. Combined hepatocellular-cholangiocarcinoma can be included.
3. HCC limited to the liver with no extra-hepatic metastasis on CT or MRI of the abdomen and chest (defined as lymph node <2 cm, lung nodules < 1 cm, farther lymph nodes < 2 cm) according to the AASLD criteria65.
4. R0 or R1 resection on histology.
5. Eligibility according to tumour size:

   1. Large tumour >= 5 cm (preferred)
   2. Smaller tumours >=2cm and < 5cm
   3. Multifocal tumours - maximum of 3 total tumours with size >=2cm detected from CT-scan. Detection of <1cm tumour intra-operatively or upon histologic examination following resection can be ignored. For multiple satellite nodules (>=2cm) that are detected intraoperatively, harvest ALL satellite nodules (>/= 2cm). DNA/RNA will be extracted from cases confirmed to be HCC/hepato-cholangiocarcinoma by histology. A MAXIMUM of 3 samples with the best quality are to be used for the analysis.
6. Child-Pugh ≤ 7 points without clinical ascites before surgery.
7. ECOG performance status 0-1 before surgery.
8. Scheduled for liver resection within 6 weeks.
9. The patient has received no anti-cancer specific treatment for HCC eg. previous liver resection, loco-regional therapy (e.g. RFA, TACE, SIRT), radiotherapy, immunotherapy, chemotherapy or neo-adjuvant chemotherapy other than the planned surgery. However, patient who has received previous HCC resection more than 5 years ago is deemed to have a de-novo liver tumour and therefore can be included.
10. Adequate bone-marrow reserve, renal function and hepatic function as assessed by standard laboratory criteria:

    * Absolute neutrophil count ≥ 1.0 x 10^9/L
    * Platelet count ≥ 50 x 10^9/L
    * Haemoglobin ≥ 9.0 g/dL
    * INR ≤ 2.0
    * Serum creatinine ≤ 1.5 times the Upper Limit of Normal (ULN)
    * Albumin ≥ 2.5 g/dL
    * Total bilirubin ≤ 1.5 times the ULN
    * Alanine transaminase (ALT) ≤ 2.5 times the ULN
    * Aspartate transaminase (AST ≤ 2.5 times the ULN

Exclusion Criteria:

1. Single lesion < 2 cm at the time of tumour resection.
2. The patient has previous or concomitant malignancies at other sites, except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and highly likely to have been cured.
3. Encephalopathy
4. The patient has received a major organ allograft.
5. The patient is known to be positive for the Human Immunodeficiency Virus (HIV).
6. The patient has an uncontrolled bleeding disorder.
7. The patient has uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease or myocardial infarction) or uncontrolled arrhythmia at the time of enrolment.
8. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent, or to comply with the study procedures.
9. The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
10. The patient has received any investigational or non-registered medicinal product (drug or vaccine) within the 30 days preceding the date of enrolment, or plans to receive such a drug during the study period.
11. For female patients: the patient is pregnant or lactating.
12. Insufficient DNA/RNA for genome analysis at baseline
13. Insufficient cells for immunology analysis at baseline (Singapore sites only)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone resection of HCC with curative intent with a R0 and R1 resection margin
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Time to recurrence | From date of Complete Response (CR) to first recurrence of HCC, up to 3 years

SECONDARY OUTCOMES:
Disease-free Survival | From date of CR to first recurrence of HCC or death, due to any cause, up to 3 years
Disease-free Specific Survival | From date of CR to first recurrence of HCC or death, due to HCC, up to 3 years
Overall Survival | From diagnosis to date of death due to any cause, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Pierce Chow, MD, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (6):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- The Medical Centre, Philippines, Manila, Philippines
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- National Cancer Institute Thailand, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen J, Kaya NA, Zhang Y, Kendarsari RI, Sekar K, Lee Chong S, Seshachalam VP, Ling WH, Jin Phua CZ, Lai H, Yang H, Lu B, Lim JQ, Ma S, Chew SC, Chua KP, Santiago Alvarez JJ, Wu L, Ooi L, Yaw-Fui Chung A, Cheow PC, Kam JH, Wei-Chieh Kow A, Ganpathi IS, Bunchaliew C, Thammasiri J, Koh PS, Bee-Lan Ong D, Lim J, de Villa VH, Dela Cruz RD, Loh TJ, Wan WK, Leow WQ, Yang Y, Liu J, Skanderup AJ, Pang YH, Ting Soon GS, Madhavan K, Kiat-Hon Lim T, Bonney G, Goh BKP, Chew V, Dan YY, Toh HC, Sik-Yin Foo R, Tam WL, Zhai W, Kah-Hoe Chow P. A multimodal atlas of hepatocellular carcinoma reveals convergent evolutionary paths and 'bad apple' effect on clinical trajectory. J Hepatol. 2024 Oct;81(4):667-678. doi: 10.1016/j.jhep.2024.05.017. Epub 2024 May 21. PMID 38782118
- [Derived] Nguyen PHD, Ma S, Phua CZJ, Kaya NA, Lai HLH, Lim CJ, Lim JQ, Wasser M, Lai L, Tam WL, Lim TKH, Wan WK, Loh T, Leow WQ, Pang YH, Chan CY, Lee SY, Cheow PC, Toh HC, Ginhoux F, Iyer S, Kow AWC, Young Dan Y, Chung A, Bonney GK, Goh BKP, Albani S, Chow PKH, Zhai W, Chew V. Intratumoural immune heterogeneity as a hallmark of tumour evolution and progression in hepatocellular carcinoma. Nat Commun. 2021 Jan 11;12(1):227. doi: 10.1038/s41467-020-20171-7. PMID 33431814